CLINICAL TRIAL: NCT02209064
Title: EASe 2- an Epicardial Access Study With the EpiAccess System- A Post-market Follow up Study.
Brief Title: "EASE" Epicardial Access With the EpiAccess System
Acronym: EASE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EpiEP, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DR-002 (rev C)
Record Dates: First submitted 2014-07-29; First posted 2014-08-05 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-02

CONDITIONS: Arrhythmias, Cardiac
Keywords: Subxiphoid; Access
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EpiAccess (Other): EpiAccess will be used to gain access to the normal, non-distended pericardial space in subjects presenting with the need for pericardial access as determined by the patient's physician.
  Interventions: Device: Pericardial access

INTERVENTIONS:
Device: Pericardial access — Access to the pericardium to enable further treatments.
  Other Names: EpiAccess

SUMMARY:
Prospective non-randomized, single arm trial to further evaluate the safety and performance of EpiAccess, the study device, for gaining access to the normal, non-distended pericardial space during epicardial diagnostic or therapeutic (ablation) procedures.

DETAILED DESCRIPTION:
Prior to enrolment, patients will be evaluated on the basis of the latest available data to establish eligibility. Eligible patients will be enrolled in the study by the local principal investigator after informed consent is obtained.

As EpiAccess is only used for the access portion of electrophysiology procedures, the safety, performance and effectiveness endpoints are acute from the time of needle insertion to pericardial space access (guidewire insertion into the pericardial sac). Patients will be followed until hospital discharge. Follow-up clinical examinations will be performed in accordance with institutions' standard of care. No special tests are required for this device. Patients' completion of study will occur at the time of their hospital discharge, or earlier if patient did not complete the study.

The stop criterion for this study is: greater than 25% Serious Adverse Device Effect, as defined in this protocol, after enrolment of 10 or more patients, compared to existing data from the literature presenting epicardial access procedure results during sub-xyphoid (minimally invasive) surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years of age or older
2. Pericardial access is clinically indicated
3. Patient is willing and able to provide written informed consent

Exclusion Criteria:

1. Patient with history of cardiac or pericardial surgery in the past 6 months
2. Patient with history of chronic pericarditis
3. Myocardial infarction within 4 weeks prior to procedure
4. Class IV NYHA (New York Heart Association) heart failure symptoms
5. Cerebrovascular accident within previous 6 months
6. Known carotid artery stenosis greater than 80%
7. Presence of thrombus in the left atrium
8. Coagulopathy
9. Severe Hepatic Dysfunction or Enlargement
10. Life expectancy less than 6 months
11. BMI > 40
12. Patient is enrolled in another clinical trial
13. Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-12; Primary Completion 2015-03 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — University of Debrecen, Cardiology/Electrophysiology Department; Debrecen, Hungary
Locations (1):
- Nemocnice Na Homolka, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tedrow U, Stevenson WG. Strategies for epicardial mapping and ablation of ventricular tachycardia. J Cardiovasc Electrophysiol. 2009 Jun;20(6):710-3. doi: 10.1111/j.1540-8167.2008.01427.x. Epub 2009 Feb 2. PMID 19207780

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 25 Patients were enrolled at five sites in Europe between February 7th 2014 and March 16, 2015
Groups:
- EpiAccess: EpiAccess was used to gain access to the normal, non-distended pericardial space in subjects presenting with the need for pericardial access as determined by the patient's physician.
  Pericardial access: Access to the pericardium to enable further treatments.
Period: Overall Study
Arm/Group | EpiAccess
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | EpiAccess
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 12
Age, Continuous [Mean (Full Range); unit: years] | 61.9 [28.4 to 84.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 19
Region of Enrollment [Number; unit: participants]
  Czech Republic | 10
  Italy | 13
  France | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Whom Pericardial Access Was Achieved With the EpiAccess System
Description: EpiAccess device shall be used to access the pericardial space with measurements tracked noting if access was achieved. The percentage of patients in whom pericardial access was successful will be reported.
Time Frame: Through discharge / approx 4 days
Population: Percentage of patients in whom epicardial access was successful using the EpiAccess system. Successful access is defined as the ability to introduce a guide wire into the epicardial space.
Measure: Number; unit: percentage of patients
Arm/Group | EpiAccess
Number analyzed (Participants) | 25
percentage of patients | 100

2. Secondary Outcome: Percentage of Participants in Whom Equivalent or Better Access Was Achieved With EpiAccess System
Description: EpiAccess will provide equivalent or better access (defined as guidewire entry into the pericardial space) as compared to access with standard of care minimally invasive, subxiphoid access techniques.
Time Frame: access through procedure completion
Measure: Number; unit: percentage of patients
Arm/Group | EpiAccess
Number analyzed (Participants) | 25
percentage of patients | 100

3. Secondary Outcome: Percentage of Participants With a Pericardial Effusion of >80ml
Description: Secondary endpoint will measure whether or not there was a pericardial effusion greater than 80ml.
Time Frame: Access through discharge/approximately 4 days
Measure: Number; unit: percentage of participants
Arm/Group | EpiAccess
Number analyzed (Participants) | 25
percentage of participants | 0

4. Other Pre Specified Outcome: Number of Patients in Whom Pericardial Access Was Achieved With the EpiAccess System
Description: Number of patients in whom the EpiAccess system was equivalently able to access the pericardial space, compared with standard of care minimally invasive access techniques,documented by using intra procedure or post procedure clinician survey
Time Frame: Access through end of procedure
Measure: Number; unit: participants
Arm/Group | EpiAccess
Number analyzed (Participants) | 25
participants | 24

ADVERSE EVENTS:
Arm/Group | EpiAccess
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 3/25
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EpiAccess (N=25)
Unintended right ventricular puncture (Cardiac disorders) | 1 (1) — Right ventricular puncture without pericardial effusion due to patient anatomy and not related to use of the EpiAccess System
Pericardial Effusion (Cardiac disorders) | 1 (1) — Pericardial effusion requiring treatment not associated with use of the EpiAccess System
Acute ischemia of left superficial femoral artery (Cardiac disorders) | 1 (1) — Not device or access related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No